CLINICAL TRIAL: NCT06413992
Title: Efficacy and Safety of Camrelizumab Plus Albumin-bound Paclitaxel/Carboplatin Followed by Camrelizumab With or Without Fluzoparib Maintenance Therapy for TP-53 Mutated Recurrent or Metastatic Endometrial Cancer: A Phase II Trial
Brief Title: Camrelizumab Plus Fluzoparib for TP-53 Mutated Endometrial Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, GUANG WEN YUAN, Professor, M.D., Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAFE
Record Dates: First submitted 2024-04-23; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Endometrial Carcinoma; TP53 Mutation; Recurrent or Metastatic
Keywords: TP53-mutated, Endometrial Carcinoma,Camrelizumab, Fluzoparib
MeSH Terms: conditions — Endometrial Neoplasms; Recurrence; Neoplasm Metastasis | interventions — fluzoparib; camrelizumab; Taxes; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab with Fluzoparib as maintainance therapy (Experimental): The treatment period mainly includes:
  1. Injection of Paclitaxel (Albumin-bound) at a dose of 260mg/m^2 administered intravenously every 3 weeks as one treatment cycle, for 6 cycles.
  2. Injection of Carboplatin (AUC=5) administered intravenously every 3 weeks as one treatment cycle, for 6 cycles.
  3. Injection of Camrelizumab at a dose of 200mg administered intravenously every 3 weeks as one treatment cycle, for 6 cycles.
  4. Radiation therapy: Not mandatory.
  Maintainance therapy period mainly includes:
  1. Injection of Camrelizumab at a dose of 200mg administered intravenously every 3 weeks as one treatment cycle until disease progression, intolerable toxicity, death, or up to a maximum of 2 years.
  2. Oral administration of Fluzoparib capsules at a dose of 150mg, once in the morning and once in the evening until disease progression, intolerable toxicity, death, or up to a maximum of 2 years.
  Interventions: Drug: Fluzoparib; Drug: Camrelizumab; Drug: paclitaxel (albumin bound); Drug: Carboplatin injection; Drug: Carboplatin; Radiation: External irradiation
- Camrelizumab without Fluzoparib as maintainance therapy (Active Comparator): Treatment period mainly include:
  1. Injection of Paclitaxel (Albumin-bound) at a dose of 260mg/m^2 administered intravenously every 3 weeks as one treatment cycle, for a total of 6 cycles.
  2. Injection of Carboplatin (AUC=5) administered intravenously every 3 weeks as one treatment cycle, for a total of 6 cycles.
  3. Injection of Camrelizumab at a dose of 200mg administered intravenously every 3 weeks as one treatment cycle, for a total of 6 cycles.
  4. Radiation therapy: Not mandatory. Whether to combine radiation therapy is determined by the principal investigator based on the patient's condition. Radiation therapy includes external beam radiation and brachytherapy.
  Maintainance therapy period mainly includes:
  a) Injection of Camrelizumab at a dose of 200mg administered intravenously every 3 weeks as one treatment cycle until disease progression, intolerable toxicity, death, or up to a maximum of 2 years.
  Interventions: Drug: Camrelizumab; Drug: paclitaxel (albumin bound); Drug: Carboplatin injection; Drug: Carboplatin; Radiation: External irradiation

INTERVENTIONS:
Drug: Fluzoparib — During the maintenance phase of treatment. Oral administration of Fluzoparib capsules at a dose of 150mg（N=78 participants）, once in the morning and once in the evening until disease progression, intolerable toxicity, death, or up to a maximum of 2 years.
  Arms: Camrelizumab with Fluzoparib as maintainance therapy
Drug: Camrelizumab — During the maintenance phase of treatment. Camrelizumab, 200 mg administered intravenously every 3 weeks until disease progression, intolerable toxicity, death, or up to 2 years.
Drug: paclitaxel (albumin bound) — Paclitaxel (albumin-bound) for injection, 260 mg/m^2 administered intravenously in 3-week cycles for 6 cycles.
Drug: Carboplatin injection — AUC=5 Intravenous dosing is administered every 3 weeks for a total of 6 treatment cycles. Specific dosing cycles may be determined by the investigator
Drug: Carboplatin — AUC=5 Intravenous dosing is administered every 3 weeks for a total of 6 treatment cycles. Specific dosing cycles may be determined by the investigator
Radiation: External irradiation — Non-essential, decision to combine is made by the principal investigator based on the patient's condition.

SUMMARY:
This study is an open-label Phase II randomized controlled trial designed to evaluate the safety and efficacy of camrelizumab plus fluzoparib maintenance therapy in patients with recurrent or metastatic TP-53 mutated Endometrial Cancer. The study will also explore the prevalence of homologous recombination reficiency in Chinese patients with TP-53 mutated endometrial cancer and its therapeutic significance.

DETAILED DESCRIPTION:
The treatment of recurrent or metastatic endometrial carcinoma (R/M-EC) has entered the era of molecular marker oriented precision therapy. Meanwhile, several large multicenter Phase III RCT studies have been conducted, such as NRG-GY018, RUBY, DUO-E and AtTEnd, and suggested that chemotherapy combined with immunotherapy could significantly improve the prognosis of R/M-EC. Unfortunately, the efficacy of ICBs in Asian R/M-EC population is not obvious, with small size.

On the other hand, up to 63% of patients with R/M-EC have TP-53 gene mutations (TP53mut). And the efficacy of chemotherapy combined with immunotherapy in thse patients is controversial. In the RUBY study, TC combined with Dostarlimab reduced the risk of death in patients with TP53mut-R/M-EC by 59 percent. However, in the DUO-E study, chemotherapy combined with Durvalumab failed to improve serous -EC in 154 patients (approximately 92% TP53mut). Therefore, how to optimize the strategy of chemotherapy combined with immunotherapy in TP53mut-R/M-EC is urgently needed.

Considering TP53mut-EC patients with tumor local T-lymph Cell infiltration and PD-L1 expression were significantly higher than those of TP-53 gene wild type (TP53wt) patients. It was also suggested that ICB and PARPi had a good synergistic effect. The DUO-E study revealed the combination of Durvalumab and Olaparib maintenance therapy significantly improves the prognosis of serous EC.

Therefore, as an investigator-initiated open-label Phase II randomized controlled study, the study will include 117 patients with TP53mut-R/M-EC, and randomly divided 2:1 into experimental group and control group to evaluate the safety and efficacy of camrelizumab plus fluzoparib maintenance therapy in patients with recurrent or metastatic TP-53 mutated Endometrial Cancer. The study will also explore the prevalence of homologous recombination reficiency in Chinese patients with TP-53 mutated endometrial cancer and its therapeutic significance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Eastern Cooperative Oncology Group (ECOG) Performance Status (ECOG): 0-2. Expected survival ≥ 6 months.
* Patients with newly diagnosed International Federation of Gynecology and Obstetrics (FIGO) 2009 stage III-IV endometrial cancer or recurrent endometrial cancer after ≤ 1 line of platinum-based chemotherapy (including neoadjuvant, adjuvant, and concurrent chemotherapy). For patients who have failed platinum-based chemotherapy, a platinum-free interval of ≥ 12 months is required.
* No restriction on pathological type, abnormal p53 expression indicated by immunohistochemistry, and confirmation of TP53 gene mutation by Sanger sequencing or next-generation sequencing (NGS).
* No prior treatment with immune checkpoint blockade (ICB) or poly (ADP-ribose) polymerase inhibitor (PARPi).
* Discontinuation of previous radiation therapy, chemotherapy, or hormone therapy for at least 4 weeks.
* Adequate organ function as follows (no use of drugs containing blood components or corrective treatment with hematopoietic growth factors in the 7 days prior to randomization): Aspartate Aminotransferase (AST) and Alanine Transaminase (ALT) ≤ 2.5 times the upper limit of normal (≤ 5 times for patients with liver metastasis) and total bilirubin ≤ 1.5 times the upper limit of normal; serum creatinine ≤ 1.5 times the upper limit of normal; platelets ≥ 90,000 cells/mm3, hemoglobin ≥ 90 g/L, and neutrophils ≥ 1,500/mm3.
* Thyroid function prior to randomization: Thyroid-stimulating hormone (TSH) level ≤ 1 times the upper limit of normal, or if TSH is not within the normal range, free T4 ≤ 1 times the upper limit of normal.
* Peripheral neuropathy grade < 2 (Common Terminology Criteria for Adverse Events, CTCAE 5.0) before treatment.
* Signed informed consent and ability to provide tumor tissue samples from initial diagnosis/recurrence for homologous recombination deficiency (HRD) testing.
* Willingness to comply with clinic visits and follow-up.

Exclusion Criteria:

* Currently participating in another clinical trial or within 4 weeks since completing another clinical trial.
* Known allergy to any components of the investigational drug.
* Previous treatment with immune checkpoint inhibitors, including but not limited to other anti-PD-1 and anti-PD-L1 antibodies.
* Patients requiring the use of immunosuppressive medications.
* Previous treatment with poly (ADP-ribose) polymerase inhibitors (PARPi).
* Patients requiring systemic or absorbable topical corticosteroids at an immunosuppressive dose, or patients who have used prednisone or equivalent drugs at a dose >10 mg/day in the two weeks prior to taking the study drug.
* Patients with any active autoimmune disease or a history of autoimmune diseases, including but not limited to active hepatitis, pneumonia, uveitis, colitis (inflammatory bowel disease), pituitary inflammation, vasculitis, nephritis, hyperthyroidism, and hypothyroidism, excluding resolved childhood asthma/atopic diseases and vitiligo. Patients with intermittent use of bronchodilators or other medical interventions for asthma should also be excluded.
* Patients in the active infectious phase requiring antimicrobial treatment (e.g., antibiotics, antiviral drugs, antifungal drugs).
* History of immunodeficiency, including human immunodeficiency virus (HIV) seropositivity or other acquired or congenital immunodeficiency diseases.
* Uncontrolled clinically significant cardiac symptoms or diseases within the past year, including but not limited to New York Heart Association (NYHA) class II or higher heart failure, unstable angina, myocardial infarction within the past year, atrial fibrillation, clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention, PR interval >250 ms, or QTc ≥470 ms.
* Arterial or venous thrombosis within the past 6 months.
* Poorly controlled hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg) despite antihypertensive medication, proteinuria ≥(++) and 24-hour total urinary protein >1.0 g.
* Coagulation abnormalities (international normalized ratio [INR] >2.0, prothrombin time [PT] >16s), bleeding tendency, or receiving thrombolytic or anticoagulant therapy.
* Patients with other malignant tumors within the past 5 years, excluding basal cell carcinoma of the skin and squamous cell carcinoma of the skin.
* Vaccination with live vaccines within 4 weeks prior to the first administration of the investigational drug. Note: Administration of inactivated seasonal influenza vaccines is allowed.
* History of substance abuse with psychotropic drugs and unable to quit, or patients with psychiatric disorders.
* The investigator believes that any other medical, psychiatric, or social factors may affect the rights, safety, ability to sign informed consent, patient's completion of the study, or interpretation of study results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed progression-free survival (PFS) | 12 months
  The time between randomization and tumor progression or death

SECONDARY OUTCOMES:
Duration of Response（DoR） | 12 months
  The duration of remission or complete disappearance of the patient's disease after treatment
Overall Survival(OS) | 24 months
  The time between randomization and death.

OTHER OUTCOMES:
Effect of HRD status and HRR-mutated on PFS | 12 months
  PFS in patients with different (Homologous Recombination Deficiency)HRD status and (Homologous Recombination Repair)HRR mutations

CONTACTS AND LOCATIONS:
Overall Officials: GUANGWEN YUAN, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No